CLINICAL TRIAL: NCT00626964
Title: Prevention of Coronary Heart Disease in Morbidly Obese Patients. Lifestyle Intervention, Low Energy Diet or Bariatric Surgery.
Brief Title: Prevention of Coronary Heart Disease in Morbidly Obese Patients
Acronym: SphCor
Status: Active, not recruiting | Type: Observational
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jøran Hjelmesæth, Professor, The Hospital of Vestfold
Other Study IDs: S-0517
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Morbid Obesity; Hypertension; Type 2 DM; Obstructive Sleep Apnea; Osteoarthrosis
Keywords: Arterial stiffness; PulseWave velocity; Body composition; Bioimpedance; Morbid Obesity; APO A; APO B; Framingham risk score; Prevention of Coronary Heart Disease; Lifestyle Intervention; Bariatric Surgery; Low Energy Diet
MeSH Terms: conditions — Obesity, Morbid; Hypertension; Sleep Apnea, Obstructive; Osteoarthritis | interventions — Bariatric Surgery; Conservative Treatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to biobank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lifestyle or bariatric surgery: Morbid Obesity with BMI >= 40 kg/m2 or BMI >= 35 with Comorbidity
  Interventions: Procedure: Bariatric Surgery; Behavioral: Conservative Treatment:

INTERVENTIONS:
Procedure: Bariatric Surgery — Bariatric Surgery Treatment: Duodenal Switch, Gastric Sleeve or Gastric bypass.
Behavioral: Conservative Treatment: — Intensive Lifestyle Intervention Program
  Other Names: Conservative

SUMMARY:
The changes in risks of developing coronary heart disease in patients with morbid obesity after different weight loss interventions have not been extensively studied. The primary objective of this study is to investigate whether an intensive lifestyle intervention program in a tertiary care clinic (Spesialsykehuset for Rehabilitering) is comparable with a 7-week low-energy-diet followed by bariatric surgery in decreasing the risk of cardiovascular disease in these patients.

DETAILED DESCRIPTION:
Patients matching the eligibility criteria were divided into two groups (not randomized). One group underwent a 7 weeks Low-Energy-Diet before bariatric surgery, the other group participated in an intensive lifestyle intervention program for 3 months.

Data on arterial stiffness, body weight, body composition, blood pressure, blood samples, vital parameters are registered in the both groups at baseline, 7 weeks and after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly Obese patients with BMI > 40, or BMI > 35 with comorbidity such as Hypertension, Obstructive Sleep Apnea, Weight Related Osteoarthrosis, Type 2 DM.

Exclusion Criteria:

* Participation in other weight loss program the last 12 months. Serious psychiatric conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly Obese patients with BMI > 40, or BMI > 35 with comorbidity such as Hypertension, Obstructive Sleep Apnea, Weight Related Osteoarthrosis, Type 2 DM.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | 7 weeks and 1 year
  Pulse wave velocity and augmentation index
Cardiovascular risk factors | 7 weeks and 1 year
  Several biomarkers will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, Principal Investigator — Morbid Obesity Center, Vestfold Hospital Trust
Locations (1):
- Morbid Obesity Center, Vestfold Hospital Trust, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young J, Seeberg KA, Aakre KM, Borgeraas H, Nordstrand N, Wisloff T, Hjelmesaeth J, Omland T, Hertel JK. The liver-heart axis in patients with severe obesity: The association between liver fibrosis and chronic myocardial injury may be explained by shared risk factors of cardiovascular disease. Clin Biochem. 2024 Jan;123:110688. doi: 10.1016/j.clinbiochem.2023.110688. Epub 2023 Nov 22. PMID 37995847
- [Derived] Berk KA, Borgeraas H, Narverud I, Mulder MT, Oyri LKL, Verhoeven AJM, Smastuen MC, Bogsrud MP, Omland T, Hertel JK, Gjevestad E, Nordstrand N, Holven KB, Hjelmesaeth J. Differential effects of bariatric surgery and lifestyle interventions on plasma levels of Lp(a) and fatty acids. Lipids Health Dis. 2022 Dec 28;21(1):145. doi: 10.1186/s12944-022-01756-1. PMID 36577984
- [Derived] Nordstrand N, Gjevestad E, Dinh KN, Hofso D, Roislien J, Saltvedt E, Os I, Hjelmesaeth J. The relationship between various measures of obesity and arterial stiffness in morbidly obese patients. BMC Cardiovasc Disord. 2011 Feb 1;11:7. doi: 10.1186/1471-2261-11-7. PMID 21284837